CLINICAL TRIAL: NCT06015880
Title: A Phase 1 Study of Mosunetuzumab With Polatuzumab Vedotin and Lenalidomide (M+Pola+Len) in Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Testing the Combination of Anti-cancer Drugs Mosunetuzumab, Polatuzumab Vedotin, and Lenalidomide for the Treatment of Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Amendment pending for dose expansion
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-06477; NCI-2023-06477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-141; 10601 (Other: City of Hope Comprehensive Cancer Center LAO); 10601 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2023-08-26; First posted 2023-08-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma; Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Specimen Handling; Lenalidomide; polatuzumab vedotin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (mosunetuzumab, polatuzumab vedotin, lenalidomide) (Experimental): Patients receive mosunetuzumab IV over 2-4 hours on days 1, 8, and 15 of cycle 1 and then day 1 of each subsequent cycle. Treatment repeats every 28 days for 8 cycles in patients who achieve a CR or up to 17 cycles for patients with a PR or SD in the absence of disease progression or unacceptable toxicity. Patients also receive polatuzumab vedotin IV over 30-90 minutes on day 1 for 6 cycles and lenalidomide PO on days 1-21 for 8 cycles in patients who achieve CR or up to 17 cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo PET/CT and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lenalidomide; Biological: Mosunetuzumab; Drug: Polatuzumab Vedotin; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Biological: Mosunetuzumab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody BTCT4465A; BTCT 4465A; BTCT-4465A; BTCT4465A; CD20/CD3 BiMAb BTCT4465A; Lunsumio; Mosunetuzumab-axgb; RG 7828; RG-7828; RG7828; RO7030816
Drug: Polatuzumab Vedotin — Given IV
  Other Names: ADC DCDS4501A; Antibody-Drug Conjugate DCDS4501A; DCDS4501A; FCU 2711; FCU-2711; FCU2711; polatuzumab vedotin-piiq; Polivy; RG 7596; RG-7596; RG7596; Ro 5541077-000
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial studies the side effects and best dose of mosunetuzumab when given together with polatuzumab vedotin and lenalidomide in treating patients with diffuse large B-cell lymphoma (DLBCL) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Mosunetuzumab and polatuzumab vedotin are monoclonal antibodies that may interfere with the ability of cancer cells to grow and spread. Polatuzumab, linked to a toxic agent called vedotin, attaches to CD79B positive cancer cells in a targeted way and delivers vedotin to kill them. Lenalidomide may stimulate or suppress the immune system in different ways and stop cancer cells from growing and by preventing the growth of new blood vessels that cancer cells need to grow. Giving mosunetuzumab with polatuzumab vedotin and lenalidomide may work better in treating patients with relapsed/refractory DLBCL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of mosunetuzumab + polatuzumab vedotin + lenalidomide in relapsed/refractory (R/R) diffuse large B cell lymphoma (DLBCL).

SECONDARY OBJECTIVE:

I. To observe and record anti-tumor activity of the combination of mosunetuzumab, polatuzumab vedotin, and lenalidomide in R/R DLBCL.

EXPLORATORY OBJECTIVES:

I. To assess the efficacy in patients that have failed prior polatuzumab vedotin containing regimens (i.e., patients who progressed/relapsed after prior polatuzumab).

II. To assess anti-tumor activity in patients that a) have < complete response (CR) or Deauville score of 3 or worse at day 90 (D90) (or before) after standard of care chimeric antigen receptor (CAR) T-cell therapy; b) other patients who have failed prior treatment (e.g. relapse after day 90 from CAR-T, or relapsed after other therapies and were not considered candidates for CAR-T).

III. To identify biomarkers that can predict the response to mosunetuzumab + polatuzumab vedotin + lenalidomide.

IV. To describe anti-tumor activity in patients whose tumors have previously failed to respond to polatuzumab (i.e., patients who progressed/relapsed after prior polatuzumab).

OUTLINE: This is a dose-escalation study of mosunetuzumab, followed by a dose-expansion study.

Patients receive mosunetuzumab intravenously (IV) over 2-4 hours on days 1, 8, and 15 of cycle 1 and then day 1 of each subsequent cycle. Treatment repeats every 28 days for 8 cycles in patients who achieve a complete response (CR) or up to 17 cycles for patients with a partial response (PR) or stable disease (SD) in the absence of disease progression or unacceptable toxicity. Patients also receive polatuzumab vedotin IV over 30-90 minutes on day 1 for 6 cycles and lenalidomide orally (PO) on days 1-21 for 8 cycles in patients who achieve CR or up to 17 cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo positron emission tomography (PET)/ computed tomography (CT) and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed DLBCL NOS, high-grade B-cell lymphoma, or transformed indolent lymphoma as per the World Health Organization 2022 criteria
* All patients will have relapsed/refractory DLBCL after 1 or more prior lines of therapy with the exception of patients receiving CAR T in second line that have a D score of 3 at day (D)+ 30 through D+ 90
* Patients who progressed/relapsed after prior polatuzumab vedotin are allowed
* For the expansion cohorts only: cohort A must have < complete response (CR) or Deauville score of 3 or 4 at D90 (or before) after standard of care chimeric antigen receptor (CAR) T-cell therapy; cohort B- other patients with relapsed/refractory after 1 or more prior lines of therapy (e.g. relapse after day 90 from CAR-T, or relapsed after other therapies and were not considered candidates for CAR-T or autologous hematopoietic cell transplantation)
* All patients that have failed 1 line of therapy will be eligible with the exception of a 12 patient cohort (A) that will require prior CAR T therapy
* Measurable disease by CT or PET scan, with one or more sites of disease >= 1.5 cm in longest dimension
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of mosunetuzumab in combination with polatuzumab vedotin, and lenalidomide in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy >= 12 weeks
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 50,000/mcL without transfusion for 2 weeks prior to cycle 1 day 1 (C1D1)
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 × institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 × ULN may be enrolled)
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 3 × ULN (AST and/or ALT =< 5 × ULN for patients with liver involvement)
* Alkaline phosphatase =< 2.5 × ULN (=< 5 × ULN for patients with documented liver involvement or bone metastases)
* Creatinine clearance >= 30 mL/min/1.73 m^2 by Cockcroft-Gault: (140- age) × (weight in kg) × (0.85 if female) 72 × (serum creatinine in mg/dL)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 × ULN (This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose.)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated

  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging 6-8 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression or CNS lymphoma
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs, as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of 1% per year during the treatment period and for 3 months after the final dose of mosunetuzumab, 3 months after the final dose of polatuzumab vedotin, and 1 month after the last dose of lenalidomide
  * For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:
  * With female partners of childbearing potential, men must remain abstinent or use a condom during the treatment period, 5 months after the final dose of polatuzumab vedotin, and 1 month after the last dose of lenalidomide
* Some concurrent cancer therapeutics (e.g., prostate, breast hormonal-based therapy) are allowed
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* Agree to comply with all local requirements of the lenalidomide risk minimization plan

Exclusion Criteria:

* Plasmablastic lymphoma, primary mediastinal B-cell lymphoma, gray zone lymphoma
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents or treatments
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to mosunetuzumab or other agents used in study
* Patients with uncontrolled intercurrent illness
* Uncontrolled or known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to first study treatment administration
* Active CNS involvement or detectable disease by lymphoma, including leptomeningeal involvement
* Pregnant women are excluded from this study because mosunetuzumab is bispecific antibody with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with mosunetuzumab, breastfeeding should be discontinued if the mother is treated with mosunetuzumab. These potential risks may also apply to other agents used in this study. Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of mosunetuzumab, 3 months after the final dose of polatuzumab vedotin, and 1 month after the final dose of lenalidomide
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2 or better
* Known or suspected chronic active Epstein-Barr virus (EBV) infection
* Patients with any other significant condition(s) that would make this protocol unreasonably hazardous

  * Current > grade 1 peripheral neuropathy
  * Prior solid organ transplantation
  * Patients with known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
  * Patients with history of confirmed progressive multifocal leukoencephalopathy (PML)
  * Currently active or uncontrolled autoimmune disease

    * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
    * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
    * Patients with a history of disease-related immune thrombocytopenic purpura, autoimmune hemolytic anemia, or other stable autoimmune diseases may be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of monsunetuzumab+polatuzumab vedotin+lenalidomide for determination of recommended phase 2 dose | During cycle 1 (cycle=28 days)
  Dose limiting toxicity will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Objective response rate | Up to 2 years
  Will be assessed per the Lugano 2014 criteria.
Complete response rate | Up to 2 years
  Will be assessed per the Lugano 2014 criteria.
Progression free survival | Up to 2 years
  Will be assessed per the Lugano 2014 criteria.
Duration of response | From time of initial response assessment demonstrating at least partial response until disease response assessment that demonstrates progressive disease, assessed up to 2 years
  Will be assessed per the Lugano 2014 criteria.

OTHER OUTCOMES:
CD79b expression levels | At baseline
  Will be assessed via ribonucleic acid and immunohistochemistry assessment and correlation with response.
Frequency of CD4 T-cells and IFN-gamma+ producing CD4 T-cells | At baseline and up to 2 years
  Will be assessed via intracellular flow cytometry.
Ultrasensitive determination of cytokine profile | At baseline and up to 2 years
  Will be assessed with Luminex assay to identify biomarkers that might predict a response.
Efficacy in relapsed/refractory double-expresser lymphoma and double-hit lymphoma | Up to 2 years
Efficacy post chimeric antigen receptor (CAR) T-cell therapy | Up to 2 years
Efficacy post polatuzumab vedotin | Up to 2 years
Percent of patients able to start the triplet therapy | At cycle 2 (cycle=28 days)
Chimeric antigen receptor (CAR) T-cell expansion and persistence | Up to 2 years
CAR T-cell immunophenotypes | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Tuscano, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm